CLINICAL TRIAL: NCT07018128
Title: Expression of Genes Relating Hypertension in Thailand and the Efficacy of 4-7-8 Breathing Control on Reducing Blood Pressure in Individuals With Hypertension
Brief Title: Expression of Genes Relating Hypertension and Efficacy of 4-7-8 Breathing Control on Reducing Blood Pressure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Burapha University (Other)
Responsible Party: Principal Investigator, Piyapong Prasertsri, Associate Professor Dr., Burapha University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB1-046/2568
Record Dates: First submitted 2025-06-01; First posted 2025-06-12 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Genetic Predisposition to Disease; Breathing, Mouth
Keywords: Gene; Blood pressure; Breathing
MeSH Terms: conditions — Genetic Predisposition to Disease; Mouth Breathing; Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: Study 1 is a cross-sectional study model and study 2 is an experimental study model.
Who Masked: Outcomes Assessor
Masking Description: Other than investigators, data collectors, and outcome adjudicators, different researchers were assigned as outcomes assessors and data analysts.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Study 2: control group (No Intervention): Participants will not receive any breathing training.
- Study 2: deep breathing (Active Comparator): Participants will practice deep diaphragmatic breathing at a rate of 6-10 breaths per minute for 15 minutes, twice a day. Participants are required to follow their assigned breathing programs daily for three consecutive months.
  Interventions: Other: Study 2: deep breathing
- Study 2: 4-7-8 breathing (Experimental): Participants will practice the 4-7-8 breathing technique, which involves inhaling for 4 seconds, holding the breath for 7 seconds, and exhaling for 8 seconds-this constitutes one cycle. They will repeat this for 6 cycles per set, three sets per day, with normal breathing between sets. Participants are required to follow their assigned breathing programs daily for three consecutive months.
  Interventions: Other: Study 2: 4-7-8 breathing
- Study 2: slow breathing with device (Active Comparator): Participants will practice deep breathing using a resistance-based breathing device called "BreathMax" which provides water pressure resistance set at 25% of their maximum inspiratory capacity. The breathing rate will be set at 6 breaths per minute, continued for 15 minutes per session, twice daily. Participants are required to follow their assigned breathing programs daily for three consecutive months.
  Interventions: Other: Study 2: slow breathing with device

INTERVENTIONS:
Other: Study 2: deep breathing — Participants in the deep breathing group will be randomized to receive a diaphragmatic deep breathing program. They will be instructed to practice deep breathing at a rate of 6-10 breaths per minute for 15 minutes, twice daily, every day for a duration of 3 months.
  Arms: Study 2: deep breathing
Other: Study 2: 4-7-8 breathing — Participants in the 4-7-8 breathing group will be randomized to receive a 4-7-8 breathing program. They will follow the 4-7-8 breathing training program, which involves inhaling for 4 seconds, holding the breath for 7 seconds, and exhaling for 8 seconds, counted as one cycle. This pattern is to be repeated for 6 cycles to complete one set. They will perform 12 sets per day-6 sets in the morning and 6 sets in the evening-with normal breathing between each set. This routine will be carried out daily for a duration of 3 months.
  Arms: Study 2: 4-7-8 breathing
Other: Study 2: slow breathing with device — Participants in the slow breathing with device group will be randomized to receive a slow breathing with device. They will undergo deep breathing training using a resistance-based breathing device called BreathMax, set at 25% of their maximal inspiratory pressure. The breathing rate will be 6 breaths per minute, continuously for 15 minutes, twice a day. This routine will be performed daily for a duration of 3 months.
  Arms: Study 2: slow breathing with device

SUMMARY:
This study consists of two sub-studies. Study 1 investigates gene expression related to the development of hypertension in Thailand, and Study 2 examines the effectiveness of the 4-7-8 breathing technique in reducing blood pressure in individuals with hypertension.

DETAILED DESCRIPTION:
In Study 1, the sample group includes 200 individuals aged 18-59 years, originating from various regions of Thailand but currently residing in the eastern region. Participants may have normal blood pressure, high blood pressure, or have been diagnosed with hypertension. Blood samples from the participants will be analyzed for the following variables: 1) expression of five genes-adrenomedullin (ADM), angiopoietin-like 4 (ANGPTL4), proto-oncogene c-Fos (FOS), prostaglandin-endoperoxide synthase 2 (PTGS2), and ubiquitin specific peptidase 8 (USP8), and 2) markers of inflammation-tumor necrosis factor-alpha and interferon-gamma levels in the blood.

In Study 2, the sample group includes 75 volunteers from Study 1 who are interested in participating. These volunteers will be randomly assigned into three groups of 25 people each. The first group is a control group whose participants will not receive any breathing training. The second group will practice the 4-7-8 breathing technique, which involves inhaling for 4 seconds, holding the breath for 7 seconds, and exhaling for 8 seconds-this constitutes one cycle. They will repeat this for 6 cycles per set, three sets per day, with normal breathing between sets. The third group will practice deep diaphragmatic breathing at a rate of 6-10 breaths per minute for 15 minutes, twice a day. Participants in both the second and third groups are required to follow their assigned breathing programs daily for three consecutive months. At the end of the three months, all participants will be assessed on the same variables measured before the intervention: 1) systolic and diastolic blood pressure levels, 2) blood pressure variability, and 3) inflammation markers, specifically tumor necrosis factor-alpha and interferon-gamma levels in the blood.

ELIGIBILITY:
Study 1:

1. Group of individuals with hypertension

   Inclusion Criteria:
   * Male or female
   * Aged between 18-59 years
   * Of Thai ethnicity
   * Diagnosed with hypertension, defined as having an SBP of 140 mmHg or higher, or a DBP of 90 mmHg or higher, or having previously been diagnosed with hypertension and currently taking antihypertensive medication
   * Originally from various regions of Thailand and currently residing in the eastern region

   Exclusion Criteria:
   * Has heart disease, such as valvular stenosis or regurgitation, coronary artery disease, or heart failure
   * Has obesity, defined as having a body mass index (BMI) of 30 kg/m² or higher
   * Has a fever or is currently experiencing an infectious disease, such as COVID-19, the flu, or other infections
2. Group of individuals with normal blood pressure

Inclusion Criteria:

* Male or female
* Aged between 18-59 years
* Of Thai ethnicity
* Does not have hypertension, defined as having an SBP below 130 mmHg and a DBP below 85 mmHg, with no prior diagnosis of hypertension and no history of taking antihypertensive medication
* Originally from various regions of Thailand and currently residing in the eastern region

Exclusion Criteria:

* Has heart disease, such as valvular stenosis or regurgitation, coronary artery disease, or heart failure
* Has obesity, defined as having a body mass index (BMI) of 30 kg/m² or higher
* Has a fever or is currently experiencing an infectious disease, such as COVID-19, the flu, or other infections

Study 2:

Inclusion Criteria:

* Male or female, aged 35-59 years
* Diagnosed with hypertension, with blood pressure levels above the normal range, defined as SBP of 130 mmHg or higher, or DBP of 85 mmHg or higher, and currently taking medication
* Originally from various regions of Thailand and currently residing in the eastern region
* Able to communicate effectively

Exclusion Criteria:

* Has respiratory diseases, cardiovascular diseases, cerebrovascular disease, kidney disease, cancer, or immune-related conditions such as allergies, autoimmune diseases (e.g., SLE), immunodeficiency, or rheumatoid arthritis
* Is obese, defined as having a body mass index (BMI) of 30 kg/m² or higher
* Has a fever or is currently infected, such as with COVID-19, the flu, or other infectious diseases
* Is currently pregnant, breastfeeding, or has a history of pregnancy within the 6 months prior to participating in the study

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Study 1: expression of adrenomedullin (ADM) | Day 1
  Expression of gene adrenomedullin (ADM) in fold unit
Study 1: expression of angiopoietin-like 4 (ANGPTL4) | Day 1
  Expression of gene angiopoietin-like 4 (ANGPTL4) in fold unit
Study 1: expression of proto-oncogene c-Fos (FOS) | Day 1
  Expression of gene proto-oncogene c-Fos (FOS) in fold unit
Study 1: expression of prostaglandin-endoperoxide synthase 2 (PTGS2) | Day 1
  Expression of gene prostaglandin-endoperoxide synthase 2 (PTGS2) in fold unit
Study 1: expression of ubiquitin specific peptidase 8 (USP8) | Day 1
  Expression of gene ubiquitin specific peptidase 8 (USP8) in fold unit
Study 1: tumor necrosis factor-alpha | Day 1
  Marker of inflammation tumor necrosis factor-alpha in picogram/milliliter unit
Study 1: interferon-gamma | Day 1
  Marker of inflammation interferon-gamma in picogram/milliliter unit
Study 2: systolic blood pressure | Day 1 and Day 85
  Systolic blood pressure in millimeter of mercury unit
Study 2: diastolic blood pressure | Day 1 and Day 85
  Diastolic blood pressure in millimeter of mercury unit
Study 2: systolic blood pressure coefficient of variation | Day 1 and Day 85
  Systolic blood pressure coefficient of variation in percentage unit
Study 2: diastolic blood pressure coefficient of variation | Day 1 and Day 85
  Diastolic blood pressure coefficient of variation in percentage unit
Study 2: tumor necrosis factor-alpha | Day 1 and Day 85
  Marker of inflammation tumor necrosis factor-alpha in picogram/milliliter unit
Study 2: interferon-gamma | Day 1 and Day 85
  Marker of inflammation interferon-gamma in picogram/milliliter unit

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Allied Health Sciences, Burapha University, MueangChonburi, Changwat Chon Buri, Thailand